CLINICAL TRIAL: NCT06204653
Title: The Effect of High-flow Nasal Oxygenation Versus Mask Ventilation on Gastric Insufflation in Children: A Randomized Controlled Trial
Brief Title: Effect of High-flow Nasal Oxygenation on Gastric Insufflation in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AJOUIRB-IV-2023-584
Record Dates: First submitted 2023-12-26; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Induction of General Anesthesia
Keywords: High flow nasal oxygenation; Facemask ventilation; Gastric insufflation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal oxygenation group (HFNO group) (Experimental)
  Interventions: Device: HFNO group
- Facemask ventilation group (MV group) (Active Comparator)
  Interventions: Device: MV group

INTERVENTIONS:
Device: HFNO group — 100% oxygen supplied in proportion to body weight using the Optiflow THRIVETM system while maintaining jaw thrust. (0-12 kg; 2 L/kg/min, 13-15 kg; 30 L/min, 16-30 kg; 35 L/min, 31-50 kg; 40 L/min)
  Other Names: Optiflow
  Arms: High-flow nasal oxygenation group (HFNO group)
Device: MV group — Mask ventilation using the one-hand E-C clamp technique and oropharyngeal airway (fresh gas flow 3 l/min, 100% O2, tidal volume 8-10 ml/kg, respiratory rate 20/min, I:E ratio 1:2, pop-off valve 13 cmH2O).
  Arms: Facemask ventilation group (MV group)

SUMMARY:
This is a randomized controlled study to compare the incidence of gastric insufflation when using high-flow nasal oxygenation and facemask ventilation in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 1 to 6 years
* American Society of Anesthesiologists physical classification 1 or 2
* Scheduled for general anesthesia

Exclusion Criteria:

* Patients expected to have difficulty with mask ventilation
* Patients with oropharyngeal facial deformity
* Obese patients (BMI>30 kg/m2)
* Patients with an upper respiratory tract infection
* Patients with a history of abdominal surgery

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of gastric insufflation | From the start of anesthesia induction to 3 minutes after anesthesia induction
  Incidence of gastric insufflation detected by gastric ultrasound (acoustic shadow phenomenon or comet-tail artifact in the antrum) or by epigastric auscultation (typical 'gurgling' or 'whoosh' sound)

SECONDARY OUTCOMES:
Gastric insufflation detected by ultrasound | 3 minutes after anesthesia induction
  Presence of acoustic shadow phenomenon or comet-tail artifact detected by ultrasound
Gastric insufflation detected by auscultation | From the start of anesthesia induction to 3 minutes after anesthesia induction
  Presence of 'gurgling' or 'whoosh' sound detected by auscultation of the epigastrium.
gastric antrum longitudinal diameter (D1) | 3 minutes after anesthesia induction
  gastric antrum longitudinal diameter (D1) measured by ultrasound
gastric antrum anteroposterior diameter (D2) | 3 minutes after anesthesia induction
  gastric antrum anteroposterior diameter (D2) measured by ultrasound
gastric antral cross-sectional area (CSA) | 3 minutes after anesthesia induction
  gastric antral cross-sectional area (CSA) measured by ultrasound (CSA = (D1 Ⅹ D2 Ⅹ π)/4)

OTHER OUTCOMES:
MAP | Every 1 minute during intervention (baseline, 1, 2, 3 min after induction)
  Mean arterial pressure
HR | Every 1 minute during intervention (baseline, 1, 2, 3 min after induction)
  Heart rate
SpO2 | Every 1 minute during intervention (baseline, 1, 2, 3 min after induction)
  Peripheral oxygen saturation
TV | Every 1 minute during intervention (1, 2, 3 min after induction)
  Tidal volume in MV group
PIP | Every 1 minute during intervention (1, 2, 3 min after induction)
  Peak airway pressure in MV group
ETCO2 | Every 1 minute during intervention (1, 2, 3 min after induction) and just after intubation
  End tidal CO2 in MV group
Lowest SpO2 | From the start of anesthesia induction to completion of tracheal intubation
  Lowest peripheral oxygen saturation during intervention